CLINICAL TRIAL: NCT05732090
Title: Effect of Diaphragmatic Myofascial Release on Thoracic Curvature Angle and Pulmonary Functions in Hyperkyphotic Adolescents
Brief Title: Effect of Diaphragmatic Myofascial Release on Thoracic Angle and Pulmonary Functions in Hyperkyphotic Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Delta University for Science and Technology (Other)
Responsible Party: Principal Investigator, Amira Hussin Hussin Mohammed, Assistant professor at faculty of physical therapy, Delta University for Science and Technology
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: diaphragm myofascial release
Record Dates: First submitted 2023-02-06; First posted 2023-02-16 (Actual); Last update posted 2024-05-22 (Actual); Status verified 2024-05

CONDITIONS: Adolescent Kyphosis
MeSH Terms: conditions — Scheuermann Disease

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (A) (Experimental): The control group will receive a therapeutic exercise program (3 sessions per week for two months).
  Interventions: Other: therapeutic exercise program
- study Group (B) (Experimental): study group will received the same intervention in control group in addition to diaphragmatic myofascial release (3 sessions/week/two months).
  Interventions: Other: therapeutic exercise program; Other: diaphragmatic myofascial release

INTERVENTIONS:
Other: therapeutic exercise program — therapeutic exercise program (3 sessions/week/two months).
Other: diaphragmatic myofascial release — therapeutic exercise program in addition to diaphragmatic myofascial release (3 sessions/week/two months).
  Arms: study Group (B)

SUMMARY:
Adolescent kyphotic girls will participate in this study. They will be divided into two groups. Group A: The control group will receive a therapeutic exercise program. Group B: The study group will receive the same intervention as Group A in addition to diaphragmatic myofascial release. They will be assessed at baseline and after three successive months of interventions for the following outcomes: Cobb angle by x-ray and pulmonary functions (vital capacity, forced vital capacity and maximum ventilatory volume) by computerized spirometer

DETAILED DESCRIPTION:
Adolescent kyphotic girls with an age range of 12-15 years old will participate in this study. They will be divided into two groups. Group A: The control group will receive a therapeutic exercise program. Group B: The study group will receive the same intervention as Group A in addition to diaphragmatic myofascial release. Both groupss will receive intervention for three three successive months. They will be be assessed at baseline and after three three successive months of interventions for the following outcomes:

Primary outcome: Cobb angle by x-ray Secondary outcome: pulmonary functions (vital capacity, forced vital capacity and maximum ventilatory volume) by computerized spirometer

ELIGIBILITY:
Inclusion Criteria:

* Adolescents girls with thoracic kyphosis with cobb angle ranged from 45 to 55 degree.
* Age ranged from 12 to 15 years old.
* selected from preparatory and secondary schools.

Exclusion Criteria:

* free from any associated deformities other than the thoracic kyphotic deformity.

Ages: 12 Years to 15 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes
Enrollment: 102 (Actual)
Dates: Start 2022-02-25 (Actual); Primary Completion 2023-05-30 (Actual); Study Completion 2023-05-30 (Actual)

PRIMARY OUTCOMES:
Cobb angle | Change from Cobb angle at 3 months
  Cobb angle by x-ray

SECONDARY OUTCOMES:
pulmonary functions (vital capacity, forced vital capacity and maximum ventilatory volume) | Change from pulmonary functions (vital capacity, forced vital capacity and maximum ventilatory volume) at 2 months
  pulmonary functions (vital capacity, forced vital capacity and maximum ventilatory volume) by computerized spirometer

CONTACTS AND LOCATIONS:
Locations (1):
- Amira Hussin Mohammed, Gamasa, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Elabd OM, Elsamahy SA, Abdelmutilibe SM, Mohammed AH, Ali F, Elabd AM. Effect of Adding Diaphragmatic Myofascial Release to Corrective Exercise on the Thoracic Curvature Angle and Pulmonary Function Testing in Hyperkyphotic Adolescent Girls: A Randomized Controlled Trial. Am J Phys Med Rehabil. 2025 Mar 1;104(3):203-209. doi: 10.1097/PHM.0000000000002622. Epub 2024 Sep 16. PMID 39331044